CLINICAL TRIAL: NCT04409951
Title: Impact of Covid-19 on Pharmacist Student Education in Egypt
Brief Title: Pharmacy Education During Covid-19 Outbreak
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Other Study IDs: Educational process & Covid-19
Record Dates: First submitted 2020-05-22; First posted 2020-06-01 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-05

CONDITIONS: Event, Life Change

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus disease 2019 (COVID-19) outbreak is considered one of the most important public health crisis all over the world. General recommendations and rules around the world have been legislated to avoid or delay transmission of covid-19. Education process and learning plan are changed to focus on online Learning instead of traditional educational model. Pharmacy is one of the important practical medical science which affected by Covid-19 outbreak.

DETAILED DESCRIPTION:
Detailed Description:

The survey will enroll as many individuals of the Egyptian pharmacy students as possible in the survey portion of the study - The number of participates have no limitations, at least 100 participants.

The survey will be enrolled in online google form, face to face interview(this will be reduced to encourage social isolation) & semi-structured telephone interviews if possible.

The research procedures:

An online survey link will include questions regarding the effect of COVID 19 pandemic on the educational process in Egypt,and how the online learning process are affecting pharmacy students it will measure the impact on the psychological health of the students as well as their level of understanding of information.and their overall satisfaction from the e learning method of education used during the COVID 19 pandemic Face to face and semi-structured interviews if possible: For those Egyptian citizens who state that they would like to participate in an interview, a random sample will be contacted.

Inclusion Criteria:

pharmacy students

Exclusion Criteria:

non pharmacy students

ELIGIBILITY:
Inclusion Criteria:

* pharmacy students

Exclusion Criteria:

* non pharmacy students

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All grades pharmacy students in Faculty of pharmacy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Impact of Covid-19 on pharmacy Education study in Egypt | 12 months
  a survey will measure the effect of the COVID 19 pandemic on the educational process in Egypt,and how the online learning process are affecting pjarmacy students.It also measures how the change in the educational process affected the psychological health of the students as well as their level of understanding of information.and their overall satisfaction from the e learning method of education used during the COVID 19 pandemic

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhour university, Beheira, Damanhour, Egypt